CLINICAL TRIAL: NCT06775262
Title: Patients with Chronic Fatigue Complaints for Whom a Consultation Including Diagnostics Do Not Reveal a Somatic Diagnosis Atthe Internal Medicine Outpatient Clinic
Brief Title: Chronic Fatigue in the Internal Medicine Outpatient Clinic: a Mixed-methods Quantitative and Qualitative Study
Status: Recruiting | Type: Observational
Sponsor: Flevoziekenhuis (Other)
Responsible Party: Sponsor
Other Study IDs: FlevoziekenhuisNL
Record Dates: First submitted 2024-12-03; First posted 2025-01-15 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Fatigue Symptom; Fatigue; Fatigue Syndrome, Chronic
Keywords: Fatigue; Qualitative study; Quantative study; Diagnostic efficacy; Internal medicine; Interviews; Grounded theory
MeSH Terms: conditions — Fatigue; Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1) Adult patients visiting the internal medicine outpatient clinic for unexplained fatigue.: Specifically the investigators will include adult patients at the above described outpatient clinic with chronic fatigue for whom a consult including diagnostics did not bring about a somatic diagnosis. This cohort is investigated in the context of the retrospective part of this study; investigating the outcome and the efficacy of diagnostics, i.e. an ECG, blood work and a chest X-ray, in patients with fatigue symptoms.
- 2) Adult patients visiting the internal medicine outpatient clinic for unexplained fatigue.: The investigators will interview patients that have visited the internal medicine outpatient clinic for unexplained fatigue symptoms for whom a consultation including diagnostics did not bring about a somatic diagnosis. The investigators will ask these patients about their experiences shortly after visiting the clinic and 6 months after. This cohort is investigated in the context of the prospective qualitative part of this study. The interviews will have an open character, in accordance with the Grounded Theory methodization.

SUMMARY:
With this study, the investigators aim to answer the following research questions:

1. In what percentage of cases does the diagnostic process conducted during a fatigue consultation at the internal medicine outpatient clinic contribute to a somatic diagnosis?
2. What are the experiences of patients presenting with fatigue at the internal medicine outpatient clinic when a consultation, including diagnostic testing, does not lead to a diagnosis?

To address question (1), the investigators will conduct a retrospective data analysis using information from HiX, an electronic health record (EHR) system.

To answer question (2), the investigators will conduct a prospective qualitative study through interviews.

DETAILED DESCRIPTION:
Chronic fatigue is a prevalent and challenging symptom, affecting an estimated 30% of the general population in the Netherlands for periods longer than six months. Despite its frequency, only a small proportion of patients presenting with fatigue receive a somatic or psychosocial diagnosis, leaving many cases unexplained. This underscores the complexity and subjective nature of fatigue, as well as the need for better understanding and management of this condition in secondary care settings.

The aim of this study is twofold. First, it seeks to determine the effectiveness of diagnostic procedures performed during fatigue consultations at an internal medicine outpatient clinic in contributing to a somatic diagnosis. Second, it aims to explore the experiences of patients for whom these consultations, including diagnostic testing, do not lead to a definitive diagnosis.

This mixed-method study combines quantitative and qualitative approaches. A retrospective analysis of medical records will assess the proportion of fatigue consultations where diagnostics, ie. blood work, an EKG and an X-thorax, result in a somatic diagnosis. Additionally, qualitative interviews will provide insight into the experiences of patients who leave the consultation without a diagnosis. The interviews will have an open characters, based ons principles of "Grounded Theory" (a qualitative research approach that generates theories from data through iterative processes of coding, comparison, and analysis, rather than testing existing hypotheses)

The study will include adult patients referred to an internal medicine outpatient clinic for unexplained fatigue. Data collection will encompass both diagnostic outcomes and patient perceptions, with findings aimed at improving care pathways and diagnostic approaches for individuals with chronic fatigue.

The study will contribute to a deeper understanding of the diagnostic process for fatigue in secondary care and offer insights into the patient experience. This knowledge has the potential to enhance clinical practices and improve patient-centered care for individuals presenting with unexplained fatigue.

ELIGIBILITY:
Cohort 1:

Inclusion Criteria:

* Patients under 18 years of age;
* Patients lost to follow-up.

Exclusion Criteria:

* Patients at the internal medicine outpatient clinic with a referral for fatigue e.c.i.
* Patients who visited the clinic after the 1st of April 2022.

Cohort 2:

Inclusion criteria

* Patients at the internal medicine outpatient clinic with a referral for fatigue e.c.i. whose consultation did not bring about a somatic diagnosis

Exclusion criteria:

* Patients under 18 years of age;
* Patients that do not speak Dutch fluently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Almere region in Flevoland who visit Flevo Hospital Almere for a fatigue consultation. They speak Dutch and are over the age of 18. For the retrospective part of this study, the investigators will exclude patients who visited the clinic during the Covid period (before the 1st of April 2022).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Results of the blood work | The investigators will determine this retrospectively, two weeks time from the time that the patients were seen.
  The investigators will determine whether or not pathology is found on the blood work that was done in the context of the fatigue consult. The investigators will determine this on the basis of the conclusion of the internal medicine specialist: Pathology: yes/no.
Results of electrocardiogram (ECG) | The investigators will determine this retrospectively, two weeks time from the time that the patients were seen.
  The investigators will determine whether or not pathology is found on the ECG that was done in the context of the fatigue consult. The investigators will determine this on the basis of the conclusion of the cardiologist: Pathology: yes/no.
Results of chest X-ray | The investigators will determine this retrospectively, two weeks time from the time that the patients were seen.
  The investigators will determine whether or not pathology is found on the chest X-ray that was done in the context of the fatigue consult. The investigators will determine this on the basis of the conclusion of the radiologist: Pathology: yes/no.
Experiences of fatigue patients visiting an internal medicine outpatient clinic for whom consultation including diagnostics did not bring about a somatic diagnosis brought about through interviews based on Grounded Theory | The investigators will explore their experiences on two moments: 1-2 months after a consultation and 6 months after a consultation and a year after consultation.
  These are adult, dutch speaking, native patients, aged 18 to 65 years. They visited the outpatient internal medicine clinic of the Flevoziekenhuis in Almere between the 1st of November 2024 until current.

CONTACTS AND LOCATIONS:
Overall Officials: Marije Ten Wolde, MD Phd, Principal Investigator — Flevoziekenhuis
Locations (1):
- Flevoziekenhuis, Almere Stad, Flevoland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided